CLINICAL TRIAL: NCT04339569
Title: Full-body Landing Biomechanics Following Fatigue in Male Jumping Athletes With and Without a History of Patellar Tendinopathy: a Case Control Study
Brief Title: Landing Biomechanics Following Fatigue in Athletes With and Without a History of Patellar Tendinopathy
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201941506
Record Dates: First submitted 2020-03-27; First posted 2020-04-09 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2019-10

CONDITIONS: Patellar Tendinitis; Fatigue
Keywords: Biomechanics; Landing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- History of patellar tendinopathy
  Interventions: Diagnostic Test: Biomechanical analysis; Other: Fatigue protocol
- Healthy controls
  Interventions: Diagnostic Test: Biomechanical analysis; Other: Fatigue protocol

INTERVENTIONS:
Diagnostic Test: Biomechanical analysis — 3D analysis of landing manoeuvres.
Other: Fatigue protocol — A circuit of different tasks (e.g. jumping, sprinting forward and backward, side-stepping exercise) was performed to induce fatigue.

SUMMARY:
In this case-control study, two- and three-dimensional landing biomechanics, by means of lower limb joint angles and moments (opto-electronic system with synchronised force plate), will be compared between 30 male volleyball/basketball players with a history of patellar tendinopathy and 30 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* volleyball or basketball players
* male
* history of patellar tendinopathy

Exclusion Criteria:

* history of surgery of the lower extremities
* history of fractures of the lower extremities

Ages: 16 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Players from sports with repetitive jump-landing manoeuvres.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Change in landing biomechanics (kinematics and kinetics) | Immediately after fatiguing exercises
  Trunk and lower extremity joint angles and moments will be extracted with an opto-electronic system and synchronised force plate

CONTACTS AND LOCATIONS:
Locations (1):
- Vakgroep Revalidatiewetenschappen, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided